CLINICAL TRIAL: NCT06259357
Title: Prone Positioning in Neurologically Deceased Potential Organ Donors to Improve Donor Lung Function and Lung Transplant Recipient Outcomes (P-POD) Pilot Trial
Brief Title: Prone Positioning in Neurologically Deceased Potential Organ Donors to Improve Donor Lung Function and Lung Transplant Recipient Outcomes
Acronym: P-POD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lorenzo delSorbo (Other)
Responsible Party: Sponsor-Investigator, Lorenzo delSorbo, MD, Critical Care Medicine Department, Toronto General Hospital, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTO 4594
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Lung Transplant Failure
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocolized protective mechanical ventilation in prone position (Experimental)
  Interventions: Other: Protocolized protective mechanical ventilation in prone position
- Protocolized protective mechanical ventilation in supine position (No Intervention)

INTERVENTIONS:
Other: Protocolized protective mechanical ventilation in prone position — Prone Position: Study subjects randomized to the intervention group will be placed and maintained in prone position for at least 16 hours/day until the time of organ procurement or decline (typically 24-48 hours after donation consent) or the time that the lungs are declined for transplant.
  Arms: Protocolized protective mechanical ventilation in prone position

SUMMARY:
The purpose of this study is to determine the practicality of performing a future, large-scale study. The future study will look at the effect of mechanical ventilation in neurologically deceased (brain-dead) lung donors who are positioned to lay flat on their stomach (prone position), compared to donors who are positioned to lay flat on their back (supine position). The study will also look at the potential impact of prone positioning of the donor on transplant recipients of the study organs.

The investigators are doing this study because the investigators want to increase the availability of donor lungs for lung transplant. Lung transplant is a life-saving treatment for individuals with lung disease, but there are not enough donated lungs to meet demand. Researchers are looking for better ways of preventing donated lungs from becoming unsuitable for transplant. Because of this, the goal of our study is to test whether prone positioning in neurologically deceased (brain-dead) lung donors can improve donor lung function and decrease complications, potentially increasing the number of donor lungs that can be used for transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Neurological determination of death at time of study entry
3. Consent to organ donation
4. Eligible for organ donation as confirmed by Trillium Gift of Life Network Coordinator

Exclusion Criteria:

1. Open chest or abdominal wounds on the ventral body surface
2. Absolute contraindication to lung transplantation on initial eligibility screening:

   * Infection i. Positive HIV, HbsAg, Human T-lymphotropic virus-I/II test results ii. Positive West Nile Virus (WNV PCR) test results iii. Rabies diagnosis or within the last 6 months bitten by an animal proven to have rabies iv. Active endocarditis v. Active encephalitis or meningitis of unknown etiology vi. Active disseminated tuberculosis vii. Viral hemorrhagic fever including Ebola or known exposure to person with Ebola viii. COVID-19 presumptive or confirmed positive in the last 14 days
   * Malignancy i. Donors with active cancer (donors receiving chemotherapy or radiation therapy or palliative cancer care within the last 5 years); excluding skin and primary brain tumors and prostate cancers.

ii. Donors with a history of the following malignancies:

* Lung Cancer
* Choriocarcinoma
* Breast Cancer
* Colon Cancer within the last 10 years iii. Donors with active or past history of melanoma o Clinician decision that prone position is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
This pilot randomized controlled trial will assess the feasibility of conducting a future full randomized clinical trial, specifically, to determine whether donor accrual will be adequate (if we recruit 40 donors from 4 sites over 1 year) | 90 days
  The number of donors enrolled into the trial over 1 year to be placed into either prone positioning or supine positioning prior to lung transplant
To document adherence to the explicit prone positioning and mechanical ventilation protocol (if more than 80% of donors have no major protocol violations then considered adequate) | 90 days
  Number of major protocol violations, specifically:
  1. Time from donation consent to randomization > 3 hours;
  2. Time from randomization to initiation of study assigned protocol > 3 hours;
  3. Time spent in prone positioning < 50% of the total time from study consent to study termination
To document the number of those who cross over to the alternate strategy (if fewer than 10% of donors cross over to the alternate strategy, when not allowed by protocol then considered adequate) | 90 days
  The percentage of donors who cross over to the alternate strategy, when not allowed by protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada